CLINICAL TRIAL: NCT05756920
Title: A Phase 1 Randomized, A Phase 1 Randomized, Placebo Controlled, Double Blind, Two Part, Single- and Multiple-Ascending-Dose Trial to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Intravenously Administered ABL301 in Healthy Adult Participants
Brief Title: This is a Study to Evaluate the Safety, Tolerability, PK and PD of IV Administered ABL301 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ABL Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABL301-1001
Record Dates: First submitted 2023-01-20; First posted 2023-03-07 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Single Ascending Dose and Multiple Ascending Dose
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABL301 (Experimental)
  Interventions: Drug: ABL301
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABL301 — SAD: Participants will receive a single dose of ABL301 IV infusion, MAD: Participants will receive multiple doses of ABL301 IV infusion
  Arms: ABL301
Drug: Placebo — SAD: single Placebo IV infusion, MAD: multiple Placebo IV infusion
  Arms: Placebo

SUMMARY:
This is a Phase 1, FIH, randomized, double-blind, placebo-controlled study designed to assess the safety, tolerability, PK and PD after SAD and MAD in healthy adult participants.

DETAILED DESCRIPTION:
The present study is the first administration of ABL301 in humans. This study will evaluate safety and tolerability and characterize the pharmacokinetic (PK) and pharmacodynamic (PD) profile of ABL301, following IV single ascending dose (Part 1 - SAD), and multiple ascending dose (Part 2 - MAD) administrations, in healthy adult participants.

In Part 1 SAD, seven single doses are planned to be administered in an ascending manner: DL1, DL2, DL3, DL4, DL5, DL6 and DL7. Each dose level will comprise 8 participants randomly assigned in an overall 6:2 ratio (ABL301:Placebo), including 1:1 ratio for the first 2 sentinel participants and 5:1 ratio for the remaining participants, to receive a single dose of study drug or placebo, respectively.

In Part 2 MAD, three multiples doses are planned to be administered in an ascending manner: DL1, DL2 and DL3. Each dose level will comprise 10 participants randomly assigned in an overall 8:2 ratio (ABL301:Placebo)

ELIGIBILITY:
Inclusion Criteria:

* The participant is considered by the investigator to be in good health as determined by medical history, clinical laboratory test results (including urinalysis), physical and neurological examination, vital signs, and ECG.
* The participant agrees to comply with all protocol requirements.
* The participant is a healthy male or female 18 to 55 years of age, inclusive.
* The participant has body weight ≥50 kg and a BMI of 19 to 30 kg/m2, inclusive.

Exclusion Criteria:

* The participant has a history of cardiovascular disease (eg, hypertension, arrhythmia, heart failure, long QT syndrome, or other conditions/diseases causing prolongation of the QT/QTcF).
* The participant has a past medical history of clinically significant ECG abnormalities or a family history of a prolonged QT interval syndrome prior to initial dosing.
* The participant has frequent headaches and/or migraine or recurrent nausea and/or vomiting (for vomiting only: more than twice a month).
* The participant has history of malignancy including solid tumors and hematologic malignancies within 5 years prior to the screening visit (except basal cell and squamous cell carcinomas of the skin that had been completely excised and were considered cured).
* The participant has a history of clinically significant drug or food allergies, as determined by the investigator.
* (MAD only) The participant has a current psychiatric disorder, suicidal ideation in the previous 6 months (as assessed by the C SSRS), or a lifetime suicide attempt.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2022-12-31 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Day 1 to Day 113 for SAD Part and D1 to Day 169 for MAD Part
  Number of participants with AEs

SECONDARY OUTCOMES:
Assessment of pharmacokinetic(PK) parameter Cmax in serum | Day 1 to Day 113 for SAD Part and D1 to Day 169 for MAD Part
  Maximum plasma concentration observed
Assessment of pharmacokinetic(PK) parameter AUClast in serum | Day 1 to Day 113 for SAD Part and D1 to Day 169 for MAD Part
  Area under the plasma concentration versus time curve from time zero to the real time tlast
Assessment of immunogenicity | Day 1 to Day 113 for SAD Part and D1 to Day 169 for MAD Part
  Numbers of subjects with ADA(anti-drug antibody) positive
Assessment of immunogenicity | Day 1 to Day 113 for SAD Part and D1 to Day 169 for MAD Part
  Numbers of subjects with ADA(anti-drug antibody) negative
Assessment of pharmacokinetic(PK) parameter AUCtau in serum (MAD only) | D1 to Day 169 for MAD Part
  Area under the serum concentration time curve over the dosing interval

OTHER OUTCOMES:
Total alpha-synuclein in plasma | Day 1 to Day 113 for SAD Part and D1 to Day 169 for MAD Part
  Plasma samples for PD analysis of ABL301 will be collected

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
ABL Bio will not be sharing individual de-identified participant data or other relevant study documents.